CLINICAL TRIAL: NCT01869621
Title: The Relation Between Heritability and the Trough Concentration of Metformin in Plasma Under Steady-state in Twins
Brief Title: Study of Metformin Pharmacogenetics in Twins
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Tore B. Stage, MSc Pharm, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AKF-383; 2012-005179-15 (EudraCT Number)
Record Dates: First submitted 2013-05-28; First posted 2013-06-05 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental): 6 days treatment with metformin
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 6 days treatment with metformin to steady-state

SUMMARY:
The trough concentration of metformin will be examined in monozygotic and dizygotic twins. Current twin study will determine the total weight of genetics on the trough concentration of metformin.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Both twins has to be included
* Dizygotic twin pairs has to be same sex
* Informed consent given
* Healthy condition

Exclusion Criteria:

* Chronical/daily alcohol abuse
* Hypersensitivity to metformin
* Ingestion of drugs containing topiramate or x-ray contrast fluids
* For women: Positive pregnancy test/breastfeeding at the beginning of the trial. No use of safe anticonceptives

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Heritability | After 6 days of metformin treatment
  The trough concentrations of metformin in twin pairs will be used to determine the effect of heritability on metformin trough concentrations. This will give insight to the weight that genetic factors have on metformin pharmacokinetics at steady-state.

SECONDARY OUTCOMES:
Single nucleotide polymorphisms (SNPs) | After 6 days treatment with metformin
  The effect of SNPs on trough metformin concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology, Odense C, Denmark